CLINICAL TRIAL: NCT05066841
Title: Chinese Herbal Medicine Formula Combined With Inhaled Corticosteroids for the Treatment of Mild to Persistent Asthma in Children: a Randomized Double-blind Placebo-controlled Trial
Brief Title: Chinese Herbal Medicine Formula Combined With Inhaled Corticosteroids for the Treatment of Mild to Persistent Asthma in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chieh Wang, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC2-111
Record Dates: First submitted 2021-09-07; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Childhood Asthma
Keywords: childhood asthma; inhaled corticosteroids; Chinese medicine; Ma-Hsing-Kan-Shih-Tang; Liu-Jun-Zi-Tang
MeSH Terms: interventions — liu-jun-zi-tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM group (Experimental)
  Interventions: Drug: CM (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang)
- placebo group (Placebo Comparator)
  Interventions: Drug: 10% CM (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang)

INTERVENTIONS:
Drug: CM (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) — CM (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) for 12 weeks
  Arms: CM group
Drug: 10% CM (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) — 10% CM (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) and 90% starch for 12 weeks
  Arms: placebo group

SUMMARY:
The purpose of study is to provide an objective data for evaluating the efficacy and safety of Chinese medicine (CM) formula combined with inhaled corticosteroid in the treatment of asthmatic children. Investigators will recruit eighty-six mild to moderate asthmatic children aged 4-11 years old with regular ICS usage and they will be randomized into two groups in this double-blind trial. Forty-three subjects will receive CM (CM group; Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) and the other forty-three subjects will receive placebo (placebo group; 10% CM) for 12 weeks. Investigators will compare these two groups by questionnaires of Childhood Asthma Control Test (cACT), the Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF), Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ), the pulmonary function test and blood test including Complete Blood Count with Differential Count (CBC/DC), total IgE, Eosinophil Cationic Protein (ECP) and IL-4/IL-5/IL-13. Adverse events, renal and liver function test will be evaluated to investigate the safety of CM formula as well.

DETAILED DESCRIPTION:
Treating pediatric asthma has been in accordance with GINA guidelines by stepwise approach to adjust treatment for individual patient needs. However, most of the asthma controller medication nowadays is inhaled corticosteroids (ICS). Parents with steroid phobia may raise concern and fears about the potential systemic effects, leading to poor adherence to medication and worse control.

This study aims to evaluate the efficacy and safety of Chinese medicine (CM) formula combined with inhaled corticosteroid for the treatment of mild to moderate persistent asthma in children. Investigators focus on the following specific aims: Aim 1. To determine the efficacy of the CM formula (Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) compared with placebo; Aim 2. To evaluate the effects of CM formula on quality of life in these patients with pediatric asthma; Aim 3. To investigate the safety of CM formula in these patients with pediatric asthma.

Eighty-six mild to moderate asthmatic children aged 4-11 years old with regular ICS usage will be randomized into two groups in this double-blind trial. Forty-three subjects will receive CM (CM group; Ma-Hsing-Kan-Shih-Tang in combination with Liu-Jun-Zi-Tang) and the other forty-three subjects will receive placebo (placebo group; 10% CM) for 12 weeks. The evaluation including pulmonary function test, IOS, FeNO, blood test, questionnaire and asthma diary card of both two groups will be conducted during the study period. The safety of CM formula use will be investigated by recording the adverse events and renal and liver function test as well.

This study will provide an objective data for evaluating the efficacy and safety o of Chinese medicine (CM) formula combined with inhaled corticosteroid in the treatment of asthmatic children. Through the combination of Chinese and western medicine, we expect to enhance the efficacy of asthma treatment, reduce acute exacerbation and tapper the dose of inhaled corticosteroids, leading to better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* aged 4-11 years old
* GINA (Global Initiative for Asthma) guideline belong to mild to moderate asthmatic children
* regular use low dose ICS+ LABA or medium dose ICS at least one month

Exclusion Criteria:

* asthma with acute exacerbation or ever has used systemic steroids in recent one month
* psychiatric disease or behavior disorder
* ever has received Chinese herbal medicine or other traditional Chinese medicine treatment in recent two weeks

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2021-09-25 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The change of Childhood Asthma Control Test (cACT) | week 12
  cACT questionnaire is a tool to evaluate asthma symptoms

SECONDARY OUTCOMES:
The change of FEV1/FVC (%) in spirometry | week 12
  Spirometry can be used to easily evaluate pulmonary function for children older than 6 years old. Participants who are unable to perform forced expiratory maneuvers will use Impulse Oscillometry System (IOS) instead.
The change of CBC/DC | week 12
  Blood test includes , total IgE, ECP and cytokines (IL-4/IL-5/IL-13) to evaluate the immunological function.
The change of total IgE | week 12
  Blood test includes CBC/DC, total IgE, ECP and cytokines (IL-4/IL-5/IL-13) to evaluate the immunological function.
The change of the ECP | week 12
  Blood test includes CBC/DC, total IgE, ECP and cytokines (IL-4/IL-5/IL-13) to evaluate the immunological function.
The change of IL-4 | week 12
  Blood test includes CBC/DC, total IgE, ECP and cytokines (IL-4/IL-5/IL-13) to evaluate the immunological function.
The change of IL-5 | week 12
  Blood test includes CBC/DC, total IgE, ECP and cytokines (IL-4/IL-5/IL-13) to evaluate the immunological function.
The change of IL-13 | week 12
  Blood test includes CBC/DC, total IgE, ECP and cytokines (IL-4/IL-5/IL-13) to evaluate the immunological function.
The change of scores of the Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF) | week 12
  ITG-CASF is a tool to measure symptoms and disability in pediatric asthma patients
The change of scores of Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) | week 12
  PACQLQ is designed to measure the limitations and anxieties faced by caregivers of children with asthma.

OTHER OUTCOMES:
The frequency of acute exacerbation | week 12
  The frequency of acute exacerbation such as ER visit and admission will be recorded in asthma diary.
Adverse drug reaction (ADR) during study period | week 12
  ADR during study period will be recorded in asthma diary.
The change of the renal function test | week 12
  Renal function test including BUN and Creatinine will to evaluate the safety of CM usage
The change of the liver function test | week 12
  Liver function test including AST and ALT will to evaluate the safety of CM usage

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan